CLINICAL TRIAL: NCT01772433
Title: The Effect of Olive Oil Phonophoresis on Chronic Low Back Pain in Female Athletes: a Randomized Controlled Trial
Brief Title: Olive Oil Phonophoresis and Chronic Low Back
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ardabil University of Medical Sciences (Other)
Collaborators: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Shahab Bohlooli, Dr, Ardabil University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1391/7/18
Record Dates: First submitted 2013-01-15; First posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Topical Olive Oil; Phonophoresis
MeSH Terms: conditions — Low Back Pain | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phonophoresis Gel (Placebo Comparator): The Phonophoresis gel will be used as placebo
  Interventions: Drug: Phonophoresis gel
- Olive Oil (Experimental): Olive oil will be used as a replacement to phonophoresis gel in this arm
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Olive oil — Phonophoresis with Olive oil for 10 day, daily
  Arms: Olive Oil
Drug: Phonophoresis gel — Phonophoresis with base gel for 10 days, daily
  Arms: Phonophoresis Gel

SUMMARY:
This study is intended to evaluate the effect of olive oil phonophoresis on chronic law back pain in female athletes.

DETAILED DESCRIPTION:
This study will enroll 60 female patients suffering from chronic low back pain. the study will run in single blind mode that only patients will kept unaware of treatment.

The duration of treatment is 10 days. patients will be assigned randomly to olive oil or placebo group. every day, they will take phonophoresis on lower back using phonophoresis gel as placebo or olive oil as treatment for 10 day. the questionnaires will be filled in baseline visit and day 10. any side effect of drugs or technique will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Young female athletes suffering from low back pain for more than three months

Exclusion Criteria:

* Underlying systematic or visceral disease
* Specific conditions such as neoplasm and fractures, spondylolisthesis
* Previous low back surgery
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Pain Score | Change from Baseline in McGill Low Back Pain Scale at day 10
  Low back pain intensity will be measured using McGill questionnaire from 0 (no pain) to 10 (worst).

SECONDARY OUTCOMES:
Physical function | Change from Baseline in Phycical Function Scale at Day 10
  The ability of patients in doing daily activities will be measured using two qualified questionnaires

OTHER OUTCOMES:
Safety | Day 10
  Any occurrence of drug induced side effects will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Bohlooli, PhD, Principal Investigator — Department of Pharmacology, School of Medicine, Ardabil University of Medical Sciences, Ardabil, Iran
Locations (1):
- Clinic of Physiotherpay, Ardabil, Ardabil Province, Iran